CLINICAL TRIAL: NCT07150702
Title: The Effect of Close Follow-up by a Physician in Addition to a Conventional Physical Therapy Program in Patients With Low Back Pain
Brief Title: Effects of Close Follow-up on Patients With Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hüdanur Coşkun, Principal Investigator, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/05/2025;2011-KAEK-50;114
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical
Keywords: low back pain; physical therapy; mechanical low back pain; pain management
MeSH Terms: conditions — Low Back Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups: the study group and the control group. Patients in the control group will undergo a conventional physical therapy program that includes hot packs, transcutaneous electrical nerve stimulation, ultrasound, and core stabilization exercises. Patients in the study group will undergo daily close follow-up physician-patient meetings during the sessions, in addition to the conventional physical therapy program applied to the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Conventional physical therapy program (Active Comparator)
  Interventions: Other: Conventional physical therapy program
- Group 2: Conventional physical therapy program with close follow-up by a physician (Active Comparator)
  Interventions: Other: Conventional physical therapy program; Behavioral: Close follow-up by a physician

INTERVENTIONS:
Other: Conventional physical therapy program — Conventional physical therapy program that includes hot packs, transcutaneous electrical nerve stimulation, ultrasound, and core stabilization exercises
Behavioral: Close follow-up by a physician — Daily physician-patient meetings during the sessions
  Arms: Group 2: Conventional physical therapy program with close follow-up by a physician

SUMMARY:
This study will include patients aged 18-65 with subacute or chronic mechanical low back pain who apply to the Physical Medicine and Rehabilitation Clinic. The age, gender, body mass index, duration of low back pain, smoking status, and educational status of the patients included in the study will be recorded. Patients will be randomized into two groups: the study group and the control group. First, the psychosocial risk status of patients in both groups will be determined using the STarT Back Screening Tool. Then, patients in the control group will undergo a conventional physical therapy program that includes hot packs, transcutaneous electrical nerve stimulation, ultrasound, and core stabilization exercises. Patients in the study group will undergo daily close follow-up physician-patient meetings during the sessions, in addition to the conventional physical therapy program applied to the control group. Clinical assessments will be performed using the Visual Analogue Scale (VAS), Tampa Scale of Kinesiophobia, Pain Catastrophizing Scale, Beck's Depression Scale, Roland-Morris Disability Questionnaire, and Leeds Assessment of Neuropathic Symptoms and Signs. Clinical evaluations will be conducted at baseline, on Day 5 post-treatment, and at 1 month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 with subacute or chronic mechanical back pain and considered appropriate for a physical therapy program.

Exclusion Criteria:

* Patients describing inflammatory back pain
* Spondyloarthropathies and other rheumatological diseases
* History of spinal surgery
* Patients with sensory disturbances and psychiatric diagnoses
* Fibromyalgia
* Patients with malignancies
* Patients with active infectious findings
* Patients with a history of radiotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | It will be evaluated in the baseline,on Day 5 post-treatment, and at 1 month post-treatment.
  Visual Analog Scale (VAS) score ranges from 0 to 10. High scores describe more pain, and low scores describe less pain.

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia | It will be evaluated in the baseline,on Day 5 post-treatment, and at 1 month post-treatment.
  The Tampa Scale of Kinesiophobia is an assessment tool typically consisting of 17 items that evaluates how much fear or anxiety individuals experience regarding movement, exercise, or physical activity. The scale ranges from a minimum score of 0 to a maximum score of 51. Higher scores indicate greater kinesiophobia (fear of movement), while lower scores reflect less fear and anxiety.
The Pain Catastrophizing Scale | It will be evaluated in the baseline,on Day 5 post-treatment, and at 1 month post-treatment.
  The Pain Catastrophizing Scale is an assessment tool that evaluates how individuals perceive pain and the level of negative thoughts and anxiety they experience related to pain. The scale typically consists of 13 items, assessing the extent to which a person catastrophizes or experiences excessive worry about their pain. Scores range from a minimum of 0 to a maximum of 52. Higher scores indicate that the individual evaluates pain in a more negative and catastrophic manner, while lower scores suggest lower levels of anxiety and catastrophizing.
Beck Depression Inventory | It will be evaluated in the baseline,on Day 5 post-treatment, and at 1 month post-treatment.
  The Beck Depression Inventory is a widely used psychometric tool for assessing the severity of an individual's depression. The scale typically consists of 21 items, each evaluating different emotional, physical, and behavioral symptoms associated with depression. Scores range from a minimum of 0 to a maximum of 63. Higher scores indicate more severe depression symptoms, while lower scores suggest fewer or less intense depressive symptoms.
Roland-Morris Disability Questionnaire | It will be evaluated in the baseline,on Day 5 post-treatment, and at 1 month post-treatment.
  The Roland-Morris Disability Questionnaire is an assessment tool designed to evaluate the functional limitations and the impact of low back pain on an individual's daily activities. The questionnaire typically consists of 24 items, each exploring how back pain affects physical activities, functionality, and quality of life. Scores range from a minimum of 0 to a maximum of 24. Higher scores indicate greater disability and more significant limitations in daily life due to back pain, while lower scores suggest fewer functional restrictions.
Leeds Assessment of Neuropathic Symptoms and Signs | It will be evaluated in the baseline,on Day 5 post-treatment, and at 1 month post-treatment.
  The Leeds Assessment of Neuropathic Symptoms and Signs is an assessment tool designed to evaluate the symptoms of neuropathic pain and the severity of these symptoms. The scale consists of 7 items, each assessing sensory changes, pain type, and the intensity of symptoms related to neuropathic pain. Scores range from a minimum of 0 to a maximum of 24. Higher scores indicate more severe neuropathic pain symptoms, while lower scores suggest milder or no neuropathic pain symptoms.

OTHER OUTCOMES:
STarT Back Screening Tool | It will be evaluated in the baseline
  The STarT Back Screening Tool is an assessment tool used to evaluate risk factors and potential functional limitations in individuals experiencing low back pain. The scale typically consists of 9 items, each addressing psychosocial factors, pain intensity, and functional capacity related to the individual's back pain. Scores range from a minimum of 0 to a maximum of 9. Higher scores indicate more severe back pain and an increased presence of psychosocial risk factors, while lower scores suggest lower risk and fewer functional limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)